CLINICAL TRIAL: NCT02765984
Title: Relation of Implantation Site to Placental Site With or Without Cesarean Section Scar
Brief Title: Relation of Implantation Site to Placental Site
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Other Study IDs: 142
Record Dates: First submitted 2016-04-30; First posted 2016-05-09 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Placenta Implantation Site
Keywords: implantation site; placental site; Doppler

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- normal placental site: women with normal implantation site at early trimester with normal placental site
  Interventions: Device: Transvaginal ultrasound
- Low placental site: women with low implantation site at early trimester with low placental site
  Interventions: Device: Transvaginal ultrasound

INTERVENTIONS:
Device: Transvaginal ultrasound — transvaginal ultrasound done before 10 weeks gestational age measuring the distance between the lower end of the hyperechoic trophoblast ring of the gestational sac and the inner cervical os

SUMMARY:
Trans vaginal ultrasound with a partially full bladder will be done at gestational age earlier than 10 weeks to assess the site of intrauterine gestational sac to the endometrial cavity and the distance between the implantation site and the internal cervical os . Doppler assessment of the retrochorionic blood flow at the area behind the maximum chorionic tissue to detect resistance index.

ELIGIBILITY:
Inclusion Criteria:

* Single intrauterine pregnancy
* Gestational age less than 10 weeks

Exclusion Criteria:

* Any condition distorting uterine cavity as myoma, uterine anomalies.
* Absent fetal pulsations
* Any condition needing termination of early pregnancy as molar pregnancy or severe deteriorating maternal disease

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women at their early trimester with or without cesarean section scar
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Distance between the implantation site and the internal cervical os | 10 weeks to 40 weeks gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Cairo University
Locations (1):
- Ahmed Maged, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided